CLINICAL TRIAL: NCT04660097
Title: Durvalumab+ Anlotinib + Standard Chemotherapy in First-line Treatment of Extensive Small-cell Lung Cancer: a Single-arm, Single-center, Phase II Clinical Study
Brief Title: Alotinib Plus Durvalumab-Platinum-Etoposide in First-line Treatment Extensive Small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yanqiu Zhao, Head of Oncology, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXNI-DA001
Record Dates: First submitted 2020-11-12; First posted 2020-12-09 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: SCLC, Extensive Stage
Keywords: small cell lung cancer, Durvalumab
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Outcome of Durvalumab-Etoposide-platinum in untreated ES-SCLC(CASPIAN trial) (Other): The outcome of CASPIAN
  Interventions: Drug: Alotinib Plus Durvalumab-Platinum-Etoposide in First-line Treatment Extensive Small-cell Lung Cancer

INTERVENTIONS:
Drug: Alotinib Plus Durvalumab-Platinum-Etoposide in First-line Treatment Extensive Small-cell Lung Cancer — This trial is single-armed IIb stage clinical trial to study the efficacy and safety of Alotinib Plus Durvalumab-Platinum-Etoposide in First-line Treatment Extensive Small-cell Lung Cancer . We use the outcome of CASPIAN trial as control group. The primary endpoint is ORR according to the RECIST 1.1, and secondary endpoints are PFS, OS, satety and life quality.
  Other Names: Anlotinib Plus Durvalumab-Platinum-Etoposide Versus Durvalumab-Platinum-Etoposide in First-line Treatment Extensive Small-cell Lung Cancer

SUMMARY:
Small Cell Lung cancer (SCLC) is a highly aggressive tumor that accounts for about 15 percent of all lung cancer cases. SCLC disease progresses rapidly, and about 2/3 of the patients have extensive stage (ES-SCLC) at the time of diagnosis, with extremely poor prognosis. However, the overall survival (OS) of ES-SCLC patients was not significantly prolonged, with platinum combined with etoposide chemotherapy as the standard treatment. In recent years, the emergence of Immune checkpoint inhibitor (ICI) has made the treatment of ES-SCLC appear at the dawn. In Impower133 study, Atezolizumab combined with chemotherapy significantly prolonged OS(median OS 12.3 months vs 10.3 months, HR=0.70, 95%CI 0.54-0.91, P = 0.007). Durvalumab combined with chemotherapy (CASPIAN study) is the first study in 20 years in which the total survival time of ES-SCLC treated by first-line therapy is 13 months, and there is no significant increase in adverse reactions compared with chemotherapy. Therefore, in 2019, NCCN also recommended Atezolizumab or Durvalumab+ EC regimens as a category 1 preferred option for first-line treatment of ES-SCLC.

DETAILED DESCRIPTION:
Small Cell Lung cancer (SCLC) is a highly aggressive tumor that accounts for about 15 percent of all lung cancer cases. SCLC disease progresses rapidly, and about 2/3 of the patients have extensive stage (ES-SCLC) at the time of diagnosis, with extremely poor prognosis. However, the overall survival (OS) of ES-SCLC patients was not significantly prolonged, with platinum combined with etoposide chemotherapy as the standard treatment. In recent years, the emergence of Immune checkpoint inhibitor (ICI) has made the treatment of ES-SCLC appear at the dawn. In Impower133 study, Atezolizumab combined with chemotherapy significantly prolonged OS(median OS 12.3 months vs 10.3 months, HR=0.70, 95%CI 0.54-0.91, P = 0.007). Durvalumab combined with chemotherapy (CASPIAN study) is the first study in 20 years in which the total survival time of ES-SCLC treated by first-line therapy is 13 months, and there is no significant increase in adverse reactions compared with chemotherapy. Therefore, in 2019, NCCN also recommended Atezolizumab or Durvalumab+ EC regimens as a category 1 preferred option for first-line treatment of ES-SCLC.

Although THE TMB of SCLC is higher in solid tumors, the objective remission rate (ORR) of SCLC using PD-1 or PD-L1 inhibitors is slightly lower than that of non-small cell lung cancer, and frequent drug resistance becomes the bottleneck of treatment. Some recent studies have shown that anti-angiogenesis drugs can also reverse the immunosuppressive state of tumor microenvironment while anti-tumor therapy, and improve the efficacy of ICI, so as to play a synergistic role. Therefore, anti-angiogenesis therapy combined with immunotherapy is expected to be a new strategy for the treatment of SCLC. Amlotinib is a multi-target anti-angiogenic drug, which has been approved for third-line treatment of SCLC with mild adverse reactions. Anlotinib combined with Durvalumab may have a synergistic antitumor effect, but no studies have been reported so far. Therefore, on the basis of the CASPIAN research study, we designed the Durvalumab + chemotherapy + ernesto, first-line treatment for extensive stage small cell lung cancer with single arm, open, multicenter, phase II clinical research, expected in domestic five cancer center, into the group of 120 ES - SCLC patients with untreated, research Durvalumab + chemotherapy + ROM for efficacy and safety of Ann, and further explore the curative effect of predictive biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary treatment of ES-SCLC (small cell lung cancer) in male or female patients aged ≥18 and <75 years.
* The ECOG energy status is 0 or 1.
* Appropriate hematologic and terminal organ functions.

Exclusion Criteria:

* Prior to systemic treatment, the patient had a history of chest radiation therapy or planned to undergo intensive chest radiation therapy.
* Spinal cord compression not explicitly treated by surgery and/or radiation, or previously diagnosed and treated, with no evidence of clinical stabilization of >2 weeks prior to randomization. Active brain metastases (stable brain metastases may be admitted after treatment) occurred within one month prior to enrollment.
* Uncontrolled or symptomatic hypercalcemia, active tuberculosis, major cardiovascular disease.
* A history of autoimmune diseases, idiopathic pulmonary fibrosis, organized pneumonia, HIV positive, active hepatitis B, radiographic findings of tumor infiltration of the large vessels in the chest and significant pulmonary cavitation lesions, a previous history of hypertensive crisis or hypertensive encephalopathy.
* History of hemoptysis within 1 month prior to randomization (≥0.5 TSP of bright red blood per episode).
* Major surgery within 28 days or needle core biopsy or other minor surgical procedures within 7 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-05-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
A Phase II, Multicenter Study to Determine the Efficacy of Anlotinib and Durvalumab in Combination With Platinum-Based Chemotherapy for the First-Line Treatment in Patients with Extensive Disease Small-Cell Lung Cancer (SCLC) . | 24 weeks
  The primary Objective of this observational study was to evaluate the Overall Survival(OS) of Durvalumab+ chemotherapy + anlotinib regimen in first-line treatment of ES-SCLC

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiu Zhao, MS, Principal Investigator — Henan Tumor Hospital
Locations (1):
- Henan Tumor Hospital, Zhengzhou, Henan, China